CLINICAL TRIAL: NCT06189352
Title: Positive Feeding of the Preterm Infant - a Feasibility Study of a Developmental Supportive Feeding Strategy in the NICU
Brief Title: Positive Feeding of the Preterm Infant
Acronym: PoP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 551058
Record Dates: First submitted 2023-11-28; First posted 2024-01-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-03

CONDITIONS: Preterm Infant; Breast Feeding; Bottle Feeding; Enteral Feeding; Cue Based Feeding; Develomentally Supportive Care
MeSH Terms: conditions — Premature Birth; Breast Feeding; Bottle Feeding

STUDY DESIGN:
Intervention Model Description: Feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The infants will follow a feeding protocol with detailed nutritional needs, and individual supportive care interventions for enhancing oral feeding development. Parents will get counseling sessions for supporting this strategy. The protocol will follow the infant until discharge.
  Interventions: Other: Positive feeding of the preterm infant

INTERVENTIONS:
Other: Positive feeding of the preterm infant — Feeding strategy for the preterm infant with description of nutritional needs and based on the infants development and cues.

SUMMARY:
The goal of this feasibility study is to assess the feasibility to implement a feeding strategy for preterm infants.

The main questions it aims to answer are:

* Is it feasible to implement the PoP-intervention in a level 3a category Neonatal intensive care unit?
* Is the PoP-intervention acceptable for parents of preterm infants and health care personnel working in Neonatal intensive care unit?

Parents of preterm infants and health care personnel will be asked to follow a protocol of a feeding strategy based on the preterm infants development and cues throughout the NICU-stay.

DETAILED DESCRIPTION:
The parents will be recruited before or as soon as possible after birth. The intervention will start as soon as the parents have given written consent for themselves and behalf of their infant.

The intervention is developed in line with the MRC framework of developing and evaluating complex interventions in an iterative and dynamic way. The intervention will be based on parents counseling and an infant feeding protocol.

ELIGIBILITY:
Inclusion Criteria:

* gestational age of 28 weeks
* post menstrual age of 28 weeks after transition from regional hospital

Exclusion Criteria:

* diagnoses or malformations that makes eating difficult
* triplets or more
* parents not speaking/understanding Norwegian or English
* parents with challenges or special needs for follow up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates and sample criteria | Prospective over a period of 1 year
  Variables to evaluate if we can recruit appropriate participants, the time frame it takes, the eligibility criterias, the recruitment routines.
Data collection and outcome variables | Prospective over a period of 1 year
  How appropriate are the data collection procedures, the participants ability to complete the quiestionnaires, appropriatness of the amount of data collection, completion of datasets,
Acceptability | Prospective over a period of 1 year
  Evaluation of acceptability of the intervention for the participants, adherence to the study procedures, the burden for participants and the health care personnell conducting the intervention, safety and adverse events
Resources and organisation | Prospective over a period of 1 year
  Evaluation of the resources needed to conduct the study procedures, resources needed for training health care personnel or other costs related to the study

SECONDARY OUTCOMES:
Infant outcome variables | Prospective over a period of 1 year
  A pilotstudy of the intervention with focus on the infants outcomes, such as weight gain, feeding milestones, nutrition, feeding methods,

CONTACTS AND LOCATIONS:
Overall Officials: Nina M Kyno, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Vestre Viken Hospital Trust, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT06189352/Prot_000.pdf